CLINICAL TRIAL: NCT04777084
Title: A Prospective, Multi-cohort Clinical Research of Efficacy and Safety of Bispecific Anti-PD-1 / PD-L1 Antibody IBI318 Combined with Lenvatinib in the Treatment of Advanced NSCLC
Brief Title: The Efficacy and Safety of the Bispecific Anti-PD-1/PD-L1 Antibody IBI318 Combined with Lenvatinib in NSCLC.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIVE
Record Dates: First submitted 2021-02-27; First posted 2021-03-02 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (Experimental): Cohort A is evaluating the efficacy and safety of IBI318 in combined with lenvatinib in advanced NSCLC patients who had failed first-line PD-1/PD-L1 inhibitor therapy.
  Interventions: Drug: IBI318
- Cohort B (Experimental): Cohort B is the efficacy and safety of advanced NSCLC with EGFR-sensitive mutation /ALK fusion after EGFR-TKI /ALK-TKI treatment resistance.
  Interventions: Drug: IBI318
- Cohort C (Experimental): Cohort C is the efficacy and safety of first-line treatment of advanced NSCLC with negative PD-L1 expression and EGFR, ALK, and ROS1 wild-type.
  Interventions: Drug: IBI318

INTERVENTIONS:
Drug: IBI318 — IBI318, 300 mg, administered by intravenous infusion on the first day of each cycle, 1 cycle every 2 weeks (Q2W), continuous medication; lenvatinib 8 mg, orally, continued medication until disease progression, death, toxicity is intolerable, Withdrawal of informed consent, start a new anti-tumor treatment or terminate the treatment for other reasons specified in the plan, the maximum use time is 2 years.

SUMMARY:
The study is a prospective multi-cohort clinical study. Cohort A is evaluating the efficacy and safety of IBI318 in combined with lenvatinib in advanced NSCLC patients who had failed first-line PD-1/PD-L1 inhibitor therapy. Cohort B is the efficacy and safety of advanced NSCLC with EGFR-sensitive mutation /ALK fusion after EGFR-TKI /ALK-TKI treatment resistance. Cohort C is the efficacy and safety of first-line treatment of advanced NSCLC with negative PD-L1 expression and EGFR, ALK, and ROS1 wild-type. After being screened to meet the inclusion criteria, they will receive IBI318 combined with lenvatinib until the disease progresses, death, toxicity is intolerable, informed consent is withdrawn, new anti-tumor therapy is started, or the treatment is terminated for other reasons specified in the plan.

DETAILED DESCRIPTION:
The study is a prospective multi-cohort clinical study. Cohort A is evaluating the efficacy and safety of IBI318 in combined with lenvatinib in advanced NSCLC patients who had failed first-line PD-1/PD-L1 inhibitor therapy. Cohort B is the efficacy and safety of advanced NSCLC with EGFR-sensitive mutation /ALK fusion after EGFR-TKI /ALK-TKI treatment resistance. Cohort C is the efficacy and safety of first-line treatment of advanced NSCLC with negative PD-L1 expression and EGFR, ALK, and ROS1 wild-type.

After being screened to meet the inclusion criteria, they will receive IBI318 combined with lenvatinib until the disease progresses, death, toxicity is intolerable, informed consent is withdrawn, new anti-tumor therapy is started, or the treatment is terminated for other reasons specified in the plan. During the treatment, RECIST v1.1 was used for clinical tumor imaging evaluation, once every 6 weeks; after 24 weeks of medication, evaluation can be done every 8 weeks.

Subjects receiving IBI318 combined with lenvatinib have the first evidence of imaging PD according to RECIST v1.1. If the subject is clinically stable, there is no evidence of rapid imaging progress, and the investigator assesses that it can continue from the study If the patient is benefited from the drug, the subject can continue the current study treatment, and the imaging evaluation must be repeated at least 6 weeks (± 7 days) later for confirmation. If PD is confirmed by re-assessment, the subject should stop the study treatment; if PD is not confirmed, the study treatment will continue, and the assessment will be carried out at the time point of the imaging examination plan specified in the plan until the PD is confirmed by imaging.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects selected for this study must meet all of the following criteria:

  1. Sign written informed consent before implementing any trial-related procedures;
  2. Age ≥18 years old and ≤75 years old;
  3. No limit on the gender;
  4. Cohort A: histological or cytological confirmed locally advanced (IIIB-IIIC) or metastatic (stage IV) NSCLC (International Association for the Study of Lung Cancer and Joint Committee on the American Classification of Cancer, TNM Lung cancer stage 8) without EGFR gene sensitive mutations, ALK gene fusion or ROS1 gene fusion confirmed by histological specimens, Relapse after failure of first-line anti-PD-1 /PD-L1 antibody therapy, as follows:

  <!-- -->

  1. Only one anti-PD-1/PD-L1 antibody monotherapy or combination therapy is accepted in the advanced stage of the disease, and other immunotherapy is not allowed;
  2. Previous anti-PD-1/L1 antibody monotherapy or combination therapy has the best curative effect (according to RECIST 1.1 criteria) as partial remission, complete remission, or stable disease for ≥6 months (defined as within 6 months from the first medication) No disease progression has occurred);
  3. Disease progression confirmed by imaging studies occurred during or after the most recent treatment.

Cohort B: histological or cytological confirmed locally advanced (IIIB-IIIC) or metastatic (stage IV) NSCLC (International Association for the Study of Lung Cancer and Joint Committee on the American Classification of Cancer, TNM Lung cancer stage 8) with histologically confirmed EGFR-sensitive mutations or ALK fusion, Relapse after failure of anti-EGFR-TKI or ALK-TKI therapy, as follows:

In patients with EGFR-tKI sensitive mutations, the specific history of previous EGFR-TKI treatment can be one of the following:

1. There is no T790M mutation in 20 exon after the failure of previous one or two generations of EGFR-TKI (including gefitinib, erlotinib, icotinib and afatinib);
2. The 20 exon T790M mutation occurred after the treatment failure of the first or second generation EGFR-TKI monotherapy (including gefitinib, erlotinib, icotinib, and afatinib, etc.), and disease progression recurred after treatment with osimertinib or other third generation EGFR-TKI;
3. Failure of prior osimertinib or other third-generation EGFR-TKI therapy as first-line therapy (regardless of EGFR T790M mutation status);
4. Those who are allowed to receive neoadjuvant/adjuvant targeted therapy in the early stage and develop drug resistance after subsequent adjuvant targeted therapy, and their drug resistance status meets one of the three requirements of appeal.

   For patients with ALK fusion NSCLC, disease progression should occur after adequate ALK-TKI treatment, and there is no opportunity for subsequent targeted therapy.

   Cohort C: Locally advanced NSCLC that is not suitable for radical surgery or radiotherapy, or that has relapsed without systematic treatment, or that has metastasized without systematic treatment and is negative for PD-L1 expression. Patients who have previously received neoadjuvant or adjuvant therapy can also receive neoadjuvant or adjuvant therapy (but neoadjuvant or adjuvant therapy is chemotherapy/radiotherapy, not immunotherapy), and the end of neoadjuvant/adjuvant therapy should be ≥6 months after tumor progression; If the pathological type is adenocarcinoma, the absence of EGFR-sensitive mutations or ALK fusion or ROS1 fusion should be confirmed. Negative expression of PD-L1 was defined as TPS <1% using 22C3 test.

5. According to the evaluation criteria for the efficacy of solid tumors (RECIST v1.1 version), there is at least one imaging measurable lesion. The lesions located in the radiation field of the previous radiotherapy can be regarded as measurable lesions if the progress is confirmed; 6. Subjects with brain metastases asymptomatic or with stable symptoms after local treatment are allowed to be included in the group, as long as the subjects meet the following conditions:

1. There are measurable lesions outside the central nervous system;
2. no symptoms of the central nervous system or no worsening of symptoms within at least 2 weeks;
3. No need for glucocorticoid therapy, or stop glucocorticoid therapy within 7 days before the first administration, or the dosage of glucocorticoid is stable and reduced to less than 10mg/day prednisone (or equivalent dose) within 7 days before the first administration ; 7. Subjects are allowed to receive palliative radiotherapy (including craniocerebral radiotherapy for symptomatic brain metastases), but the radiotherapy must be completed at least 1 week before enrollment, and the radiotherapy-related toxicity should be restored to less than or equal to 1 degree (CTCAE 5.0, except for hair loss).

8. ECOG score 0-1 points; 9. Expected survival time> 3 months; 10. Sufficient organ function, subjects need to meet the following laboratory indicators:

1. The absolute value of neutrophils (ANC) ≥1.5x109/L when no granulocyte colony-stimulating factor is used in the past 14 days;
2. In the case of no blood transfusion in the past 14 days, platelets ≥100×109/L;
3. In the past 14 days without blood transfusion or erythropoietin, hemoglobin>9g/dL;
4. Total bilirubin≤1.5×upper limit of normal (ULN);
5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within ≤2.5×ULN (subjects with liver metastases are allowed to have ALT or AST ≤5×ULN);
6. Serum creatinine ≤1.5×ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥50ml/min;
7. Good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN;
8. Normal thyroid function is defined as thyroid-stimulating hormone (TSH) within the normal range. If the baseline TSH is out of the normal range, subjects whose total T3 (or FT3) and FT4 are within the normal range can also be included in the group;
9. Myocardial enzyme spectrum is within the normal range (for example, simple laboratory abnormalities that are judged by the investigator to be of no clinical significance are also allowed to be included in the group); 11. For female subjects of childbearing age, a urine or serum pregnancy test and the result should be negative within 3 days before receiving the first study drug administration (day 1 of cycle 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women of non-bearing age are defined as at least 1 year after menopause, or have undergone surgical sterilization or hysterectomy; 12. If there is a risk of conception, all subjects (whether male or female) need to adopt a low annual failure rate during the entire treatment period until 120 days after the last study drug administration (or 180 days after the last study drug administration) Less than 1% of contraceptive measures; 13. Blood pressure can be adequately controlled with or without anti hypertensive medication, defined as blood pressure≤150/ 90 mm Hg, and blood pressure was under stable control within 1 week before randomization.

14. Patients must have recovered from toxicity or complications if they have previously received surgery or radiation > 30Gy.

Exclusion Criteria:

* Subjects who meet the following criteria cannot be selected for this study:

  1. The pathology is small cell lung cancer (SCLC), including lung cancer mixed with SCLC and NSCLC;
  2. There is imaging evidence of tumor voids, tumor inclusion or invasion of large vessels. In addition, the proximity of the tumor to the large blood duct should be considered and the risk of severe bleeding associated with tumor shrinkage/necrosis after lenvatinib treatment should be excluded. (The large vessels in the chest include the main pulmonary artery, left pulmonary artery, right pulmonary artery, 4 pulmonary veins, superior vena cava, inferior vena cava and aorta);
  3. To cohort A: subjects who have previously used anti-PD-1, PD-L1 or other immunotherapy and meet the following conditions:

  <!-- -->

  1. The toxicity that caused permanent discontinuation occurred before the termination of immunotherapy;
  2. Prior to the administration of the study drug, the toxicity of the previous immunotherapy has not recovered or has not recovered to level 0-1. Asymptomatic and stable control of endocrine toxicity level 2 with appropriate replacement therapy is allowed to enter the group;
  3. Adverse events that require additional immunosuppressive agents in addition to corticosteroids, or adverse events that still recur in the use of corticosteroids during previous immunotherapy.

To cohort B and C: Prior treatment: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulating or co-inhibiting T-cell receptor (including but not limited to CTLA-4, OX-40, CD137, etc.); Anti-pd-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulating or co-inhibiting T cell receptor (including but not limited to CTLA-4, OX-40, CD137, etc.); 4. Have received the following treatments:

1. Received systemic anti-tumor therapy within 2 weeks before treatment, such as chemotherapy, targeted therapy, immunotherapy (including Chinese herbal medicine with anti-tumor indications), etc.;
2. Previously received lenvatinib, bevacizumab, anlotinib monotherapy, or in combination with anti-PD-1 / PD-L1 drugs
3. Have received any investigational drug treatment within 4 weeks before treatment;
4. Received large doses of immunosuppressive drugs within 4 weeks before treatment (systemic glucocorticoid exceeding 10mg/day prednisone or its equivalent dose);
5. Received live attenuated vaccine within 4 weeks before treatment (or plan to receive live attenuated vaccine during the study period);
6. Have received major surgery (such as open cavity, thoracotomy, or Kaifu surgery), or unhealed surgical wounds, ulcers or fractures within 4 weeks before treatment.

5. Clinically significant cardiovascular damage occurred within 12 months of the first dose of study treatment.

6. Gastrointestinal diseases that may affect oral absorption of study drugs. 7. Prior gastrointestinal or grade ≥3 non-gastrointestinal fistula. 8. A history of other malignancies is known, and unless the participant has undergone potentially curative treatment, there is no evidence of disease recurrence in the 3 years since the start of that treatment.

9. Severe allergy to IBI318 and lenvatinib. 10. There is clinically uncontrollable pleural effusion/abdominal effusion (subjects who do not need to drain the effusion or stop drainage for 3 days without a significant increase in effusion can be included in the group); 11. Subjects who have received thoracic radiotherapy of greater than 30 Gy within 6 months before treatment or palliative radiotherapy of 30 Gy or less within 7 days before treatment (allowing palliative treatment of bone lesions or intracranial lesions) Radiation Therapy); 12. An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, glucocorticoids, or immunosuppressive agents) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments; 13. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 14. Before starting treatment, have not fully recovered from toxicity and/or complications caused by any intervention (ie, ≤ Grade 1 or reached baseline, excluding fatigue or hair loss); 15. Known history of human immunodeficiency virus (HIV) infection (ie HIV 1/2 antibody positive); 16. Untreated active hepatitis B (defined as HBsAg positive and the number of HBV-DNA copies detected at the same time is greater than the upper limit of the normal value of the laboratory department of the research center);

Note: Hepatitis B subjects who meet the following criteria can also be included in the group:

1. Before the first administration, the HBV viral load is less than 1000 copies/ml (200 IU/ml), and the subject should receive anti-HBV treatment during the entire study chemotherapy drug treatment to avoid viral reactivation
2. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), there is no need to receive preventive anti-HBV treatment, but close monitoring of virus reactivation is required 17. Active HCV infected subjects (HCV antibody-positive and HCV-RNA level is higher than the lower limit of detection); 18. Live vaccines have been vaccinated within 30 days before the first administration (cycle 1, day 1); Note: It is allowed to receive inactivated virus vaccine for seasonal influenza injection within 30 days before the first administration; however, it is not allowed to receive live attenuated influenza vaccine for intranasal administration.

19. Pregnant or lactating women; 20. There are any serious or uncontrollable systemic diseases, such as:

1. The resting electrocardiogram has major abnormalities in rhythm, conduction or morphology that are severe and difficult to control, such as complete left bundle branch block, heart block above degree II, ventricular arrhythmia or atrial fibrillation;
2. Left ventricular ejection fraction (LVEF) was lower than normal; 3）QTc interval is extended to more than 480 ms；

4) Unstable angina pectoris, congestive heart failure, chronic heart failure of New York Heart Association (NYHA) grade ≥ 2; 5) Myocardial infarction occurred within 6 months before enrollment; 6) A history of non-infectious pneumonia requiring glucocorticoid treatment within 1 year before the first administration, or current clinically active interstitial lung disease; 7) Active tuberculosis; 8) There is an active or uncontrolled infection that requires systemic treatment; 9) There is clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction; 10) Liver diseases such as liver cirrhosis, decompensated liver disease, acute or chronic active hepatitis; 11) Poor control of diabetes (fasting blood glucose (FBG)> 10mmol/L); 12) Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein quantification is confirmed to be greater than 1.0 g; 13) Subjects who have mental disorders and cannot cooperate with treatment; 21. The medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the test results, prevent the subject from participating in the study, or the investigator believes that it is not suitable for inclusion this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
12 weeks ORR | 1 year
  Defined as the proportion of subjects achieving a complete remission (CR) or partial remission (PR) at around 12 weeks after the start of study treatment among all subjects.

SECONDARY OUTCOMES:
PFS | 1 year
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)
DCR | 1 year
  Defined as the proportion of subjects with complete remission (CR), partial remission (PR) and stable disease (SD) to the total subjects
DOR | 1 year
  Defined as the time interval from the first record of disease remission to disease progression or death (whichever occurs first)
OS | 1 year
  Defined as the time from the start of treatment to the death of the subject due to any cause.
BOR | 1 year
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects
adverse events (safety) | 1 year
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No